CLINICAL TRIAL: NCT02085226
Title: Can an Arts Based Creative Engagement Intervention Following Stroke Improve Psychosocial Outcomes? A Feasibility Trial of a Creative Engagement Intervention for In-patient Rehabilitation
Brief Title: Art as Creative Engagement for Stroke
Acronym: ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: University of Stirling (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011GM01; CZH/4/720 (Other Grant/Funding Number: Chief Scientist Office, Scotland)
Record Dates: First submitted 2014-03-06; First posted 2014-03-12 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Stroke
Keywords: Stroke; Rehabilitation; Creative Engagement; Psychosocial; Art
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creative Engagement Intervention (Experimental): Creative Engagement Intervention participants will receive 4-8 art sessions over 3-5 weeks, depending on length of inpatient stay. Sessions will be delivered as 1:1 sessions with the artist lasting up to one hour (depending on patient fatigue levels) and group sessions, with up to 5 participants, lasting up to two hours (depending on patient fatigue levels). Participant with receive one group and one individual session per week of inpatient stay. The sessions will cover 5 activity stages of the intervention, taking the participant through a progressive artwork development process. Participants will explore basic visual art materials and processes and progress to creating artworks with a personal context that they have directed and controlled.
  Interventions: Other: Creative Engagement Intervention
- Portfolio Group (Placebo Comparator): The Portfolio group will receive conventional rehabilitation activity at each site. In addition, to control for effects of art related attention received by the intervention group, after baseline assessment and randomisation, this group will receive from the research assistant, a portfolio of work produced by previous participants of the Tayside CEI, with details of community programmes that people with stroke can attend after hospital discharge. Participants will be invited to view the portfolio during their stay. Prior to outcome assessment, the research assistant will visit participants again to answer questions and to discuss options for community programmes, if the person is interested.
  Interventions: Other: Portfolio Group

INTERVENTIONS:
Other: Creative Engagement Intervention — The CEI has 5 component stages which map the participant's journey with the Artist
  1. Meeting with Artist, discuss interests, stroke and explore initial creative goals.
  2. Introduction to materials and mark making to create interpretations of established images.
  3. From mark making and interpretations to developing personal project ideas.
  4. Turning personal project ideas into creative finished pieces.
  5. Review of completed work, mounting and display of work, future plans.
  It is recognised that participants will progress differently. Components may be repeated or retuned to or may be addressed simultaneously. Participants may progress rapidly and so move from stage 5 back to stages 2, 3 or 4 to progress new work or experience new materials or processes.
  Other Names: CEI
  Arms: Creative Engagement Intervention
Other: Portfolio Group — The Portfolio group will receive conventional rehabilitation activity at each site. In addition, to control for effects of art related attention received by the intervention group, after baseline assessment and randomisation, this group will receive from the research assistant, a portfolio of work produced by previous participants of the Tayside CEI, with details of community programmes that people with stroke can attend after hospital discharge. Participants will be invited to view the portfolio during their stay. Prior to outcome assessment, the research assistant will visit participants again to answer questions and to discuss options for community programmes, if the person is interested.
  Arms: Portfolio Group

SUMMARY:
Title: A C E S Study: Can an arts based creative engagement intervention (CEI) following stroke improve psychosocial outcomes? A feasibility trial of a creative engagement intervention for inpatient rehabilitation.

This is a feasibility randomised controlled trial of a novel intervention for stroke rehabilitation examining effects of participation in visual arts activities on psychosocial outcomes after stroke.

The investigators hypothesise that participation in a visual arts based intervention (CEI) will improve stroke recovery variables, mood and self-esteem in stroke survivors receiving in-patient rehabilitation compared to viewing a portfolio of artwork.

The results of the study will inform a sample size calculation for a full trial.

DETAILED DESCRIPTION:
SUMMARY

Background: Stroke is the main cause of complex adult disability in Britain. Stroke rehabilitation is typically task orientated, focusing on physical and functional independence. Psychosocial consequences of stroke are serious and mediate recovery, influencing family relationships, community reintegration and quality of life. Therefore, improving psychosocial outcomes after stroke could improve overall recovery.

Creative arts programmes are increasingly used to address psychosocial outcomes in long-term and mental health conditions. These programmes focus on positive influences of engagement in creative art activities facilitated by artists. However, there is little research into effects of creative engagement on psychosocial outcomes after stroke.

Objectives: The purpose of this study is to:

Conduct a feasibility randomised controlled trial (RCT) to test the effects of a participatory visual arts intervention compared to art viewing on psychosocial outcomes following stroke in order to assess effect size for sample size calculation in a full RCT.

The effects of the CEI will be examined in a randomised controlled feasibility trial, which will be run at two stroke rehabilitation units in NHS Tayside and will explore the impact of the intervention on a range of psychosocial outcomes.

Patients meeting inclusion criteria will be randomised to a CEI group or an attention control group. The CEI group will receive a visual arts intervention of 4-8 sessions during in-patient rehabilitation. The control group will receive an art portfolio to view after randomisation and baseline assessment, with information about community opportunities to engage in art. The groups will be compared on selected psychosocial outcomes. Findings will indicate the potential magnitude and direction of change to allow for sample size requirements in development of a subsequent randomised control trial to examine effectiveness of the CEI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stroke
* Medically stable and referred for rehabilitation
* Able to sit upright in chair
* 3 or more weeks of rehabilitation planned

Exclusion Criteria:

* Diagnosis of Transient Ischemic Attack
* Patinet in acute medical need
* Patient unable to provide informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-07; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Stroke Impact Scale | Assessed at end of intervention at 4 weeks

SECONDARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | Assessed at end of intervention at 4 weeks
Visual Analogue Self-Esteem Scale (VASES) | Assessed at end of intervention at 4 weeks

OTHER OUTCOMES:
Trait Hope Scale | Assessed at end of intervention at 4 weeks
General Self Efficacy Scale | Assessed at end of intervention at 4 weeks
Self-Efficacy for Art Scale | Assessed at end of intervention at 4 weeks
Recovery Locus Of Control Scale (RLOC) | Assessed at end of intervention at 4 weeks
Stroke Impact Scale | 16 weeks
Positive and Negative Affect Scale | 16 weeks
Visual Analogue Self-Esteem Scale | 16 weeks
Trait Hope Scale | 16 weeks
General Self-Efficacy Scale | 16 weeks
Self-Efficacy for Art Scale | 16 weeks
Recovery Locus of Control Scale | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jacqui H Morris, PhD, Principal Investigator — University of Dundee; Brian Williams, PhD, Study Chair — University of Stirling; Thilo Kroll, PhD, Study Chair — University of Dundee; Gillian Mead, PhD, Study Chair — University of Edinburgh; Peter Donnan, PhD, Study Chair — University of Dundee
Locations (2):
- United Kingdom (2):
  - NHS (National Health Service) Tayside, Stroke Rehab Unit, Stracathro Hospital, Brechin, Angus
  - NHS Tayside, PRI Stroke Unit, Perth Royal Infirmary, Perth, Perth & Kinross

REFERENCES:
- [Background] Morris J, Toma M, Kelly C, Joice S, Kroll T, Mead G, Williams B. Social context, art making processes and creative output: a qualitative study exploring how psychosocial benefits of art participation during stroke rehabilitation occur. Disabil Rehabil. 2016;38(7):661-72. doi: 10.3109/09638288.2015.1055383. Epub 2015 Jun 18. PMID 26084571
- [Background] Morris JH, Kelly C, Toma M, Kroll T, Joice S, Mead G, Donnan P, Williams B. Feasibility study of the effects of art as a creative engagement intervention during stroke rehabilitation on improvement of psychosocial outcomes: study protocol for a single blind randomized controlled trial: the ACES study. Trials. 2014 Sep 28;15:380. doi: 10.1186/1745-6215-15-380. PMID 25262168
- [Result] Morris JH, Kelly C, Joice S, Kroll T, Mead G, Donnan P, Toma M, Williams B. Art participation for psychosocial wellbeing during stroke rehabilitation: a feasibility randomised controlled trial. Disabil Rehabil. 2019 Jan;41(1):9-18. doi: 10.1080/09638288.2017.1370499. Epub 2017 Aug 30. PMID 28853296